CLINICAL TRIAL: NCT02212574
Title: Pilot Study Assessing the Feasibility of a Surgery and Chemotherapy-Only Approach in the Upfront Therapy of Children With Wnt Positive Standard Risk Medulloblastoma
Brief Title: Study Assessing the Feasibility of a Surgery and Chemotherapy-Only in Children With Wnt Positive Medulloblastoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Participant relapses led to abrupt stop of study.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Matthew Larson Foundation for Pediatric Brain Tumors (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1403; NA_00091840 (Other: JHMIRB)
Record Dates: First submitted 2014-07-07; First posted 2014-08-08 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Medulloblastoma
Keywords: Wnt; Medulloblastoma; Chemotherapy
MeSH Terms: conditions — Medulloblastoma | interventions — Lomustine; Vincristine; Cisplatin; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Other): Chemotherapy Cycle A Lomustine (CCNU) is given by mouth on Day 1. Vincristine is given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, and 15. Cisplatin is given directly into a vein over 8 hours on Day 1. This cycle lasts 42 days.
  Chemotherapy Cycle B Cyclophosphamide is given into a vein over 1 hour on Days 1 and 2. MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 and 6 hours. Vincristine is given directly into a vein directly into the vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 and 8.This cycle lasts 28 days
  Interventions: Drug: Lomustine; Drug: Vincristine; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Mesna

INTERVENTIONS:
Drug: Lomustine — Chemotherapy Cycle A Lomustine (CCNU) is given by mouth on Day 1.
  Other Names: CCNU
Drug: Vincristine — Chemotherapy Cycle A Vincristine is given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, and 15.
  Other Names: Oncovin
Drug: Cisplatin — Chemotherapy Cycle A Cisplatin is given directly into a vein over 8 hours on Day 1.
  Other Names: Cisplatinum
Drug: Cyclophosphamide — Chemotherapy Cycle B Cyclophosphamide is given into a vein over 1 hour on Days 1 and 2.
  Other Names: Cytoxan
Drug: Mesna — Chemotherapy Cycle B MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 and 6 hours.
  Other Names: Mesnex
Drug: Vincristine — Chemotherapy Cycle B Vincristine is given directly into a vein directly into the vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 and 8.
  Other Names: Oncovin

SUMMARY:
Participants enrolling on this study will receive standard of care chemotherapy for Wnt positive medulloblastoma without the radiation therapy or the weekly chemotherapy that is given during radiation therapy.

DETAILED DESCRIPTION:
There will be 9 cycles of chemotherapy. There are two different kinds of cycles given. They are referred to as A and B.

Cycle A lasts for 6 weeks and Cycle B lasts for 4 weeks. B cycles are given after the completion of two A cycles.

Below are the details of the drugs and schedules for A and B cycles.

Cycle A (This cycle lasts 42 days)

* Lomustine (CCNU) is given by mouth on Day 1.
* Vincristine is given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, and 15.
* Cisplatin is given directly into a vein over 8 hours on Day 1

Cycle B (This cycle lasts 28 days)

* Cyclophosphamide is given into a vein over 1 hour on Days 1 and 2.
* MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 and 6 hours.
* Vincristine is given directly into a vein directly into the vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 and 8.

You may also get a supportive care drug called a myeloid growth factor (filgrastim or pegfilgrastim). This drug will help your blood counts recover after the chemotherapy is given.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have classical histology posterior fossa medulloblastoma as determined by institutional neuro-pathological evaluation.
* Sufficient pathologic material must be available for central analysis and review
* Tumors will be deemed Wnt positive if, at the time of central analysis, there is:
* Monosomy 6 as determined by array CGH
* Gene transcript detection by NanoString supporting Wnt+ medulloblastoma
* Absence of large-cell, anaplastic histology
* Nuclear b-catenin IHC will be determined, but not required for the diagnosis
* Absence of residual or disseminated disease as defined by the following criteria: Minimal residual disease as determined by post-operative imaging preferably performed within 48 hours of resection (and at most 28 days post-surgery), i.e. gross total resection or residual disease of <1.5cm2 on post-operative imaging.

No evidence of metastatic disease in the brain, spine or cerebral spinal fluid (CSF). Assessments must include MRI imaging of the brain and spine with and without contrast and a lumbar puncture for CSF cytology

* Diagnostic imaging (pre and post contrast) must be forwarded to Dana-Farber Cancer Institute (DFCI) for central review to confirm eligibility
* Patients must not have had any radiation therapy or chemotherapy for medulloblastoma prior to study enrollment
* Patients must have a Lansky performance status of >/=30 for children </=10 years of age or a Karnofsky performance status of > 30 for children > 10 years of age.
* Participants must have normal organ and marrow function as defined below:
* Hemoglobin greater than 10 g/dL (can be transfused). Hemoglobin <10 g/dL due to operative blood loss is permitted.
* Absolute neutrophil count > 1.0x109/L
* Platelets > 100,000/uL (non-transfused)
* Total bilirubin <1.5 x upper limit normal
* SGOT (AST) or SGPT (ALT) <2.5 x upper limit normal (ULN) for age
* Creatinine clearance or radioisotope GFR >70 ml/min/1.73m2 or normal serum creatinine for patient's age and gender
* All females of child-bearing age must have a negative pregnancy test before being enrolled on study. All patients of child-bearing age must practice an effective method of birth control whilst undergoing chemotherapy on study.
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, lomustine, vincristine or cyclophosphamide.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cohen, MD, Study Chair — Johns Hopkins University
Locations (16):
- United States (16):
  - Phoenix Childrens Hospital Hematology/Oncology, Phoenix, Arizona
  - Children's Hospital Colorado Center for Cancer & Blood Disorders, Aurora, Colorado
  - M D Anderson Cancer Center-Orlando Pediatric Hematology/Oncology, Orlando, Florida
  - All Children's Hospital Pediatric Hematology/Oncology, St. Petersburg, Florida
  - Children's Healthcare of Atlanta- Egleston Pediatric Neuro-Oncology, Atlanta, Georgia
  - Ann and Robert H Lurie Children's Hospital of Chicago Hematology/Oncology, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine Pediatric Hematology/Oncology, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University Pediatric Hematology/Oncology, Portland, Oregon
  - Seattle Children's Hospital Hematology/Oncology, Seattle, Washington
  - Childrens Hospital of Wisconsin (Medical College of Wisconsin), Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day 1. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15. Cisplatin given directly into a vein over 8 hours on Day 1. Cycle lasts 42 days.
  Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2. MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.Cycle lasts 28 days Lomustine: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day Vincristine: Chemotherapy Cycle A Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15.
  Cisplatin: Chemotherapy Cycle A Cisplatin given directly into a vein over 8 hours on Day 1.
  Cyclophosphamide: Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2.
  Mesna: Chemotherapy Cycle B MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours.
  Vincristine: Chemotherapy Cycle B Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.
Period: Overall Study
Arm/Group | Chemotherapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy: Chemo Cycle A Lomustine (CCNU) given by mouth on Day 1. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15. Cisplatin given directly into a vein over 8 hours on Day 1. Cycle lasts 42 days.
  Chemo Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 and 2. MESNA, a drug to protect the bladder from effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide, repeated at 3 and 6 hours. Vincristine given directly into a vein directly into the vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8. Cycle lasts 28 days Lomustine: Chemotherapy Cycle A Lomustine (CCNU) is given by mouth on Day 1. Vincristine: Chemo Cycle A Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15.
  Cisplatin: Chemo Cycle A Cisplatin is given directly into a vein over 8 hours on Day 1.
  Cyclophosphamide: Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2.
  Mesna: Chemo Cycle B MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide, repeated at 3 & 6 hours.
  Vincristine: Chemo Cycle B Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 7 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine the feasibility of treating newly diagnosed children with non-metastatic, standard risk, Wnt positive medulloblastoma with a chemotherapy-only approach. Primary outcome measure of this study will be progression-free survival; the number of participants who with progression free survival.
Time Frame: 3 years
Population: This outcome was not assessed because some patients had a relapse and study was abruptly terminated.
Groups:
- All Patients: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day 1. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15. Cisplatin given directly into a vein over 8 hours on Day 1. Cycle lasts 42 days.
  Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2. MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.Cycle lasts 28 days Lomustine: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day Vincristine: Chemotherapy Cycle A Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15.
  Cisplatin: Chemotherapy Cycle A Cisplatin given directly into a vein over 8 hours on Day 1.
  Cyclophosphamide: Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2.
  Mesna: Chemotherapy Cycle B MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours.
  Vincristine: Chemotherapy Cycle B Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Patterns of Failure
Description: To evaluate the patterns of failure in those children that do not have progressive disease, progression free survival and overall survival.
Time Frame: 3 years
Population: This outcome was not assessed because some patients had a relapse and study was abruptly terminated.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events were not collected for standard of care chemotherapy.
Groups:
- All Participants: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day 1. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15. Cisplatin given directly into a vein over 8 hours on Day 1. Cycle lasts 42 days.
  Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2. MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours. Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.Cycle lasts 28 days Lomustine: Chemotherapy Cycle A Lomustine (CCNU) given by mouth on Day Vincristine: Chemotherapy Cycle A Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1, 8, & 15.
  Cisplatin: Chemotherapy Cycle A Cisplatin given directly into a vein over 8 hours on Day 1.
  Cyclophosphamide: Chemotherapy Cycle B Cyclophosphamide given into a vein over 1 hour on Days 1 & 2.
  Mesna: Chemotherapy Cycle B MESNA, a drug to protect the bladder from the effects of cyclophosphamide, will be given 15 minutes before each dose of cyclophosphamide and repeated at 3 & 6 hours.
  Vincristine: Chemotherapy Cycle B Vincristine given directly into a vein (IV) over one minute or using a minibag over several minutes by some institutions on Days 1 & 8.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Two of the participants relapsed not long into the study and the Data and Safety Management Committee (DSMC) recommended early closure of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02212574/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02212574/SAP_001.pdf
  • Informed Consent Form (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT02212574/ICF_002.pdf